CLINICAL TRIAL: NCT02892851
Title: A Pilot Study of Deep Brain Stimulation of the Sub-thalamic Nucleus to Treat Treatment-resistant Cocaine Addiction With Severe Somatic or Psychiatric Complications
Brief Title: Deep Brain Stimulation of the Sub-Thalamic Nucleus to Treat Severe and Treatment-resistant Cocaine Addiction.
Acronym: STUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P111014
Record Dates: First submitted 2016-08-18; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Cocaine Addiction
Keywords: STN-DBS; Craving; Cocaine addiction
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep brain stimulation (DBS) (Experimental): Deep brain stimulation of the subthalamic nuclei (STN-DBS)
  Interventions: Device: Deep brain stimulation of the subthalamic nuclei (STN-DBS)

INTERVENTIONS:
Device: Deep brain stimulation of the subthalamic nuclei (STN-DBS) — 3 phases :
  * Parameter setting
  * Cross-over double-bind (ON/OFF)
  * Open Phase (ON)
  Other Names: Activa PC Medtronic (7428) stimulator

SUMMARY:
Cocaine addiction is a chronic condition with severe cardiac, neurologic, psychiatric and social complications. Cocaine is the second most consumed illicit drug in France. Its prevalence has been multiplied by 3 between 2000 and 2008, and is still on the rise. Craving, the compulsive need to consume, is a key feature of cocaine addiction. It is also predictive of treatment efficacy. However, there is no validated treatment for severe cocaine dependence yet. Response to current psychological and medical treatment is poor, with 73% relapse after 3 months. Patients with severe cocaine addiction are thus in a therapeutic deadlock.

To address these unmet medical needs, the investigators designed a pilot study (n=2) to evaluate the safety and the efficacy of the deep brain stimulation of the subthalamic nuclei (STN-DBS) in severe cocaine addiction with at least one cardiac, neurologic or psychiatric complication. Indeed, compulsivity is a critical component of craving, and severe treatment-resistant obsessive compulsive disorder (OCD) are already successfully treated using STN-DBS. Moreover, animal studies recently demonstrated a therapeutic effect of STN-DBS in rats addicted to cocaine. Together, these two lines of research suggest a therapeutic effect of STN-DBS in cocaine addiction mediated by an anti-obsessive mechanism on craving.

ELIGIBILITY:
Inclusion Criteria:

* severe and resistant Cocaine Dependence for 5 years defined as:

  * cocaine dependence (DSM IV),
  * preferential use of cocaine in base form (crack or free-base) through smoke,
  * non response to at least two well-conducted treatment with at least a stay in aftercare,
  * severe physical complications (defined as a history of myocardial infarction, stroke).
* psychotic syndromes induced recurrent, severe lung disease "crack-lungs") occurred due to crack consumption and whose association with the crack use is known to the patient
* age between 30 and 55 years
* patient affiliated to a social security scheme
* patient signed an informed consent after receiving written information on the proposed procedure

Exclusion Criteria:

* a current opioid dependence will not be a criterion of non inclusion if the patient is undergoing substitution treatment (methadone or buprenorphine) and not injection of opiates for at least six months.
* patient trust
* pregnant, nursing or of childbearing potential without effective contraception
* current use of the intravenous route for the administration of the drugs is the risk of infection
* VIH infection or VHC unstabilized,
* cardiovascular and / or brain state is not compatible with the surgery,
* other disorder on Axis I not linked to cocaine use except:

  * current or past dependence to nicotine,
  * abuse or dependence on other psychoactive substances over a lifetime in remission for more than 6 months,
  * current opioid dependence: if the patient is undergoing substitution treatment (methadone or buprenorphine) and not injection of opiates for at least 6 months,
  * when other psychiatric disorders induced by substances.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Evolution of the Obsessive Compulsive Cocaine Scale (OCCS) craving score | at month 6

SECONDARY OUTCOMES:
Psychiatric assessment by standardized interview | Month -2, Month 2, Month 3, Month 3+15 days, Month 4+15days, Month 6, Month 7, Month 8, Month 9, Month10 (+1,5)
Cocaine Craving Questionnaire (CCQ) craving score | Month -2, Month 2 (1day), Month 2 (2nd day), Month 2 (3rd day), Month 3, Month 3+15 days, Month 4+15days, Month 6, Month 7, Month 8, Month 9, Month 10 (+1,5)
Self assessed addiction criteria | Month -2, Month 2, Month 3, Month 3+15 days, Month 4+15days, Month 6, Month 7, Month 8, Month 9, Month10 (+1,5)
Urine screening assay for cocaine use / Urine Drug Screening | Month -2, Month 2, Month 3, Month 3+15 days, Month 4+15days, Month 6, Month 7, Month 8, Month 9, Month10 (+1,5)
Capillary screening assay for cocaine use | Month -2, Month 4,5 and Month 10 (+1,5)
Evolution of Global Assessment of Functioning scale (GAF) | Month -2, Month 2, Month 3, Month 3+15 days, Month 4+15days, Month 6, Month 7, Month 8, Month 9, Month10 (+1,5)

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No